CLINICAL TRIAL: NCT00988650
Title: Mechanistic Investigation of the Mediterranean Diet and Its Impact on the Metabolic Syndrome in Men
Brief Title: Mediterranean Diet and the Metabolic Syndrome
Acronym: MedDiet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Benoit Lamarche, Professor, Laval University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: INAF-2006-277
Record Dates: First submitted 2009-09-25; First posted 2009-10-02 (Estimated); Last update posted 2013-03-05 (Estimated); Status verified 2013-03

CONDITIONS: Cardiovascular Disease
Keywords: Metabolic syndrome; Mediterranean diet; Blood lipids; Coronary heart disease; Apolipoprotein
MeSH Terms: conditions — Cardiovascular Diseases; Metabolic Syndrome; Coronary Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- North American diet (Active Comparator): Control North American diet for five weeks in isocaloric conditions
  Interventions: Other: isocaloric diet
- Mediterranean diet (Experimental): Mediterranean diet for five weeks in isocaloric conditions
  Interventions: Other: isocaloric diet
- weight loss period (Experimental): Weight loss period of 20-week (minimum 5% reduction in body weight)
  Interventions: Other: free living conditions
- Weight stabilizing mediterranean diet (Active Comparator): Mediterranean diet for five weeks in isocaloric weight stabilizing conditions
  Interventions: Other: isocaloric diet

INTERVENTIONS:
Other: isocaloric diet
  Other Names: 3 isocaloric die
  Arms: Mediterranean diet; North American diet; Weight stabilizing mediterranean diet
Other: free living conditions
  Other Names: weight lost free living conditions
  Arms: weight loss period

SUMMARY:
While there is now undisputable evidence relating elevated plasma low-density lipoprotein (LDL) cholesterol levels to an increased risk of coronary heart disease (CHD), it is being increasingly recognized that a significant proportion of CHD events occur in individuals characterized by a cluster of additional metabolic and physiological perturbations now defined as the metabolic syndrome. Epidemiological and clinical evidence have shown us that nutritional factors, often in conjunction with obesity, play a pivotal role in the pathophysiology of the metabolic syndrome. In that regard, accumulating evidence suggest that a Mediterranean-style diet (MedDiet) may beneficially modify several components of the metabolic syndrome including plasma triglycerides (TG) and high-density lipoprotein (HDL) cholesterol levels, insulin resistance, waist circumference and markers of vascular inflammation. However, the physiological mechanisms underlying the cardioprotective effects of the MedDiet on features of the metabolic syndrome and the importance of body weight reduction in maximizing these effects represent key issues that have yet to be investigated.

The general objective of the study is to investigate for the first time in a controlled feeding study the mechanisms and factors underlying the impact of the MedDiet, with and without weight loss on the dyslipidemic features of the metabolic syndrome.

DETAILED DESCRIPTION:
The study has a duration of 35 weeks for each participant. Subjects will be first assigned to a North American control diet that they will consume for five weeks under isocaloric, weight-maintaining conditions. Participants will then consume the MedDiet for 5 weeks, again under isocaloric, weight-maintaining conditions. All foods will be provided to participants during these consecutive 5-week diets. Participants subsequently will then undergo a 20-week weight loss period in free-living conditions during which they will be given advice on how to create a 500 kcal deficit in their daily energy intake. The last phase of the study consists of a second 5-week MedDiet consumed under feeding, weight stabilizing conditions. Metabolic studies and CHD risk factor assessment will be performed at the end of each experimental diets. Metabolic studies include the measurement of in vivo kinetics of apolipoprotein (apo)B-containing lipoproteins including small dense LDL, apoCIII, HDL (apoAI) and C-reactive protein (CRP) as well as indirect measures of cholesterol absorption and synthesis.

ELIGIBILITY:
Inclusion Criteria:

* Men from the Québec City metropolitan area with the metabolic syndrome based on the NCEP-ATP III definition (3 criteria or more see below):
* Waist circumference ≥ 102 cm
* Triglycerides ≥ 1.7 mmol/L
* HDL-cholesterol <= 1.04 mmol/L
* Systolic blood pressure ≥ 130 mmHg or diastolic blood pressure ≥ 85 mmHg
* Fasting blood glucose ≥ 5.6 mmol/L
* Stable body weight (+/- 2 kg) for 6 months before the beginning of the study

Exclusion Criteria:

* Previous history of cardiovascular disease, type 2 diabetes and monogenic dyslipidemia
* Subjects taking medications for hyperlipidemia or hypertension
* Endocrine disorders
* Food allergies or aversion for specific components of the MedDiet
* Smokers
* Consummation excessive of alcohol (> 2 consummation/day)

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2007-05; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
plasma LDL, TG and HDL-C | Week 5, 10 and 35 (at the end of each weight-maintaining diet)

SECONDARY OUTCOMES:
CRP, and blood pressure, kinetic of lipoproteins | Week 5, 10 and 35 (at the end of each weight-maintaining diet)

CONTACTS AND LOCATIONS:
Overall Officials: Benoît Lamarche, PhD, Study Director — Institute of Nutraceutical and Functional Foods (INAF), Laval University
Locations (1):
- Institute of Nutraceutical and Functional Foods (INAF), Laval University, Québec, Quebec, Canada

REFERENCES:
- [Derived] Richard C, Couture P, Desroches S, Nehme B, Bourassa S, Droit A, Lamarche B. Effect of an isoenergetic traditional Mediterranean diet on the high-density lipoprotein proteome in men with the metabolic syndrome. J Nutrigenet Nutrigenomics. 2014;7(1):48-60. doi: 10.1159/000363137. Epub 2014 Jul 4. PMID 25011605
- [Derived] Richard C, Couture P, Desroches S, Lichtenstein AH, Lamarche B. Effect of an isoenergetic traditional Mediterranean diet on apolipoprotein A-I kinetic in men with metabolic syndrome. Nutr J. 2013 Jun 7;12(1):76. doi: 10.1186/1475-2891-12-76. PMID 24499022
- [Derived] Richard C, Couture P, Ooi EM, Tremblay AJ, Desroches S, Charest A, Lichtenstein AH, Lamarche B. Effect of Mediterranean diet with and without weight loss on apolipoprotein B100 metabolism in men with metabolic syndrome. Arterioscler Thromb Vasc Biol. 2014 Feb;34(2):433-8. doi: 10.1161/ATVBAHA.113.302185. Epub 2013 Nov 21. PMID 24265415
- [Derived] Richard C, Couture P, Desroches S, Lamarche B. Effect of the Mediterranean diet with and without weight loss on markers of inflammation in men with metabolic syndrome. Obesity (Silver Spring). 2013 Jan;21(1):51-7. doi: 10.1002/oby.20239. PMID 23505168